CLINICAL TRIAL: NCT03448107
Title: Comparative Effectiveness of Treatments to Prevent Dental Caries Given to Rural Children in School-based Settings: Protocol for a Cluster Randomized Controlled Trial
Brief Title: Comparative Effectiveness of Treatments to Prevent Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU College of Dentistry (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Richard Niederman, Professor, NYU College of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: i17-01221; R01MD011526 (NIH)
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries
Keywords: dental caries; caries arrest; caries prevention; silver diamine fluoride; sealants; interim therapeutic restorations
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, non-inferiority cluster randomized trial
Who Masked: Outcomes Assessor
Masking Description: The investigators responsible for analyzing the data for primary outcomes will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Simple Prevention (Experimental): One drop (0.05 ml) of silver diamine fluoride (Advantage ArrestTM) solution at 38% concentration (2.24 F-ion mg/dose) will be dispensed per child. Posterior tooth surfaces to be treated will be dried, after which the SDF will be applied with a micro-brush to all asymptomatic carious lesions and to all pits and fissures on bicuspids and molar teeth for thirty seconds. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Interventions: Device: Silver Diamine Fluoride; Device: Fluoride Varnishes
- Complex Prevention (Active Comparator): Pits and fissures on all bicuspids and molar teeth will be sealed with glass ionomer sealants (GC Fuji IX). Glass ionomer sealants (interim therapeutic restorations) will also be placed on all frank asymptomatic carious lesions. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Interventions: Device: Fluoride Varnishes; Device: Glass Ionomer

INTERVENTIONS:
Device: Silver Diamine Fluoride — Silver diamine fluoride (SDF)
  Other Names: Advantage Arrest
  Arms: Simple Prevention
Device: Fluoride Varnishes — Fluoride varnish (FV)
Device: Glass Ionomer — Glass Ionomer Sealants (GC Fuji IX)
  Arms: Complex Prevention

SUMMARY:
Dental caries (tooth decay) is the most prevalent childhood disease in the world. Multiple interventions are available to treat and prevent caries. The aim of the proposed study is to compare the benefit of silver diamine fluoride (SDF) and fluoride varnish versus fluoride varnish and glass ionomer sealants. This study is a five-year, cluster randomized, pragmatic controlled trial conducted in public elementary schools in New Hampshire.

DETAILED DESCRIPTION:
Dental caries is the most prevalent childhood disease in the world and can lead to infection, pain, reduced quality of life, and negative educational outcomes. Multiple prevention agents are available to arrest and prevent dental caries, however little is known of the comparative effectiveness of combined treatments in pragmatic settings. The aim of the presented study is to compare the benefit of silver diamine fluoride and fluoride varnish versus fluoride varnish and glass ionomer therapeutic sealants in the arrest and prevention of dental caries.

This is a longitudinal, pragmatic, cluster randomized, single-blind, non-inferiority trial to be conducted in low-income children enrolled in public elementary schools in New Hampshire from 2017-2023. The primary objective is to assess the non-inferiority of alternative agents in the arrest and prevention of dental caries. Caries arrest will be evaluated after two years, and caries prevention will be assessed at the completion of the study. Data analysis will follow intent to treat, and statistical analyses will be conducted using a two-sided significance level of 0.05.

Notably, the standard of care for dental caries is office-based surgery, which presents multiple barriers to care including cost, fear, and geographic isolation. The simplicity and affordability of silver diamine fluoride may be a viable alternative for the arrest and prevention of dental caries in high-risk children.

ELIGIBILITY:
Inclusion Criteria:

* Any primary school with a previously employed caries prevention program operating in rural areas, with official Title 1 status, and located in a health professional shortage area. Within participating schools, all children are eligible to participate in the study. Those with informed consent and assent will receive care.

Exclusion Criteria:

* Children without informed consent or those with consent but without assent.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3345 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Niederman, DMD, Principal Investigator — NYU Langone Health; Ryan R Ruff, MPH, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University College of Dentistry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data could be shared with proper approval from participating organizations for relevant and appropriate requests.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available December 1, 2025 and for five years.
Access Criteria: By request of the original principal investigators.

REFERENCES:
- [Derived] Ruff RR, Niederman R. School-based caries prevention using silver diamine fluoride: A pragmatic randomized trial in low-income rural children. medRxiv [Preprint]. 2024 Jun 25:2024.06.05.24308499. doi: 10.1101/2024.06.05.24308499. PMID 38883737
- [Derived] Ruff RR, Niederman R. Comparative effectiveness of treatments to prevent dental caries given to rural children in school-based settings: protocol for a cluster randomised controlled trial. BMJ Open. 2018 Apr 13;8(4):e022646. doi: 10.1136/bmjopen-2018-022646. PMID 29654053

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Groups:
- Simple Prevention: One drop (0.05 ml) of silver diamine fluoride (Advantage ArrestTM) solution at 38% concentration (2.24 F-ion mg/dose) will be dispensed per child. Posterior tooth surfaces to be treated will be dried, after which the SDF will be applied with a micro-brush to all asymptomatic carious lesions and to all pits and fissures on bicuspids and molar teeth for thirty seconds. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Silver Diamine Fluoride: Silver diamine fluoride (SDF)
  Fluoride Varnishes: Fluoride varnish (FV)
- Complex Prevention: Pits and fissures on all bicuspids and molar teeth will be sealed with glass ionomer sealants (GC Fuji IX). Glass ionomer sealants (interim therapeutic restorations/atraumatic restorations) will also be placed on all frank asymptomatic carious lesions. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Fluoride Varnishes: Fluoride varnish (FV)
  Glass Ionomer: Glass Ionomer Sealants (GC Fuji IX)
Period: Overall Study
Arm/Group | Simple Prevention | Complex Prevention
Started | 1558; 17 Schools | 1787; 18 Schools
Completed | 1329; 17 Schools | 1529; 18 Schools
Not Completed | 229; 0 Schools | 258; 0 Schools
Not completed — Lost to Follow-up | 229 | 258

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simple Prevention | Complex Prevention | Total
Number analyzed (Participants) | 1558 | 1787 | 3345
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (1.8) | 7.3 (1.8) | 7.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 784 | 808 | 1592
  Male | 774 | 979 | 1753
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 13 | 23 | 36
  Black | 16 | 14 | 30
  White | 346 | 522 | 868
  Asian | 10 | 19 | 29
  Multiple | 10 | 9 | 19
  Other | 1 | 9 | 10
  Unreported | 1162 | 1191 | 2353
Baseline untreated decay [Count of Participants; unit: Participants] | 221 | 276 | 497

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Arrested Dental Caries, Assessed Using a Clinical Oral Examination
Description: For any participants with untreated dental caries on teeth at baseline treated with SDF/FV or Glass ionomer atraumatic restorative treatment (ART)/FV to arrest (control) the infection, what is the proportion of participants that stayed arrested
Time Frame: Two years
Population: The analysis population are those participants who completed the study and had dental caries at baseline. This population is a subset of the full study population.
Measure: Count of Participants; unit: Participants
Arm/Group | Simple Prevention | Complex Prevention
Number analyzed (Participants) | 115 | 157
Participants | 48 | 53

2. Primary Outcome: Caries Prevention
Description: For teeth without carious lesions (sound teeth) treated with SDF/FV or Glass ionomer/FV, how many teeth developed caries over the course of observation
Time Frame: Five years
Population: The analysis population includes the total number of teeth in each participant in each group. Thus, the overall number of units analyzed will be greater than the number in participant flow (participant flow reflects individuals participating in the study).
Measure: Number; unit: teeth
Units Other Than Participants: Teeth
Arm/Group | Simple Prevention | Complex Prevention
Number analyzed (Participants) | 543 | 540
Number analyzed (Teeth) | 10860 | 10800
teeth | 210 | 179

ADVERSE EVENTS:
Time Frame: Study participants were monitored for adverse events through study completion (5 years, 8 months; average per-participant duration 2.2 years).
Arm/Group | Simple Prevention | Complex Prevention
All-Cause Mortality (participants affected / at risk) | 0/1558 | 0/1787
Serious Adverse Events (participants affected / at risk) | 0/1558 | 0/1787
Other Adverse Events (participants affected / at risk) | 0/1558 | 0/1787

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03448107/Prot_SAP_001.pdf